CLINICAL TRIAL: NCT00397436
Title: Pilot Study of Protein Profiling of the Human Epidermal Cells After Ultraviolet Irradiation
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0506M70827
Record Dates: First submitted 2006-11-07; First posted 2006-11-09 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Proteomics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Comparing irradiated skin to non irradiated skin.
  Interventions: Procedure: UV Irradiation

INTERVENTIONS:
Procedure: UV Irradiation — UV irradiation
  Other Names: UV irradiation.

SUMMARY:
The main focus of this pilot study is to construct a fairly complete protein profile of the epidermis. This will allow us to study how the epidermis responds to external stressors such as ultra-violet. We hypothesize that by using the cutting edge technology, proteomics, we will be able to construct a fairly complete profile of different epidermal cells (keratinocytes, epidermal nerve fibers (ENFs), melanocytes, Langerhans cell,...etc) of normal and ultraviolet (UV) irradiated skin.

DETAILED DESCRIPTION:
We will investigate the changes of the epidermal cell proteome after UV irradiation to the forearms of healthy young male volunteers. Knowledge of specific molecular markers may provide knowledge of basic biological systems and possibly targeted therapy of inflammation.

By using combined proteomic methodologies we will be able to quantify protein changes at cytoplasmic and membrane protein levels of epidermal cells in normal vs. irradiated skins.

This study may allow us to obtain fairly comprehensive profile of membrane integrated and cytoplasmic proteins of epidermal cell populations which will facilitate our understand of biological responses to UV irradiation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Males age 18-30
* Caucasian
* No neurological disease

Exclusion Criteria:

* Use of any medication that affects skin

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2007-02; Primary Completion 2011-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Ability to quantify protein changes at cytoplasmic and membrane protein levels of epidermal cells in normal vs. irradiated skin | 1 year

SECONDARY OUTCOMES:
Obtain a profile of membrane integrated and cytoplasmic proteins of epidermal cell populations which will facilitate our understanding of biological responses to UV irradiation. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: George Wilcox, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States